CLINICAL TRIAL: NCT06349824
Title: Dextrose, Steroid, PRP: Choosing the Right Injection for Long Term CRS Relief; a RCT
Brief Title: Dextrose, Steroid, PRP: Choosing the Right Injection for CRS Relief; a RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Sairah Sadaf, Assistant professor, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 004AEstb/EC/01/2022
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dextrose (Experimental)
  Interventions: Device: USG machine
- Steroid (Experimental)
  Interventions: Drug: injection Dextrose water; Device: USG machine
- PRP (Experimental)
  Interventions: Drug: injection Dextrose water; Device: USG machine

INTERVENTIONS:
Drug: injection Dextrose water — dextrose will be injected around median nerve in wrist
  Other Names: PRP
  Arms: PRP; Steroid
Device: USG machine — usg guided nerve hydrdissection

SUMMARY:
USG guided injections to relieve carpal tunnel syndrome with dextrose water or steroid or PRP

ELIGIBILITY:
Inclusion Criteria:

* NA

Exclusion Criteria:

* Na

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
VAS | five to six months
  visual pain score at different intervals

CONTACTS AND LOCATIONS:
Overall Officials: sairah sadaf, Principal Investigator — sheikh zayed medical college rhaim yar khan
Locations (1):
- Sheikh Zayed Medical College, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided